CLINICAL TRIAL: NCT06185452
Title: Implementation of Out-of-HOspital Administration of the Long-Acting Combination Cabotegravir+Rilpivirine as an Optional Therapy in HIV-Infected Patients From Spain: Acceptability, Appropriateness, Feasibility and Satisfaction: The HOLA Study
Brief Title: Implementation of Out-of-HOspital Administration of the Long-Acting Cabotegravir+Rilpivirine
Acronym: HOLA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Out-of-hospital LA CAB+RPV
Record Dates: First submitted 2023-09-22; First posted 2023-12-29 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; long acting; primary center; community center; out-of-hospital by implementation; cabotegravir + rilpivirine (CAB+RPV)
MeSH Terms: interventions — cabotegravir; Rilpivirine; Organization and Administration

STUDY DESIGN:
Intervention Model Description: A 12-months prospective, hybrid type (implementation-effectiveness), phase IV, randomized (1:1), open label, multicentric study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hospital Group (Active Comparator): Administration of long-acting Vocabria (cabotegravir) 600 mg and long-acting Rekambys (rilpivirine) 900 mg in the hospital (standard of care)
  Interventions: Drug: Hospital long-acting Vocabria (cabotegravir) 600 mg and long-acting Rekambys (rilpivirine) 900 mg administration
- Outpatient Group (Experimental): Out-of-hospital administration of long-acting Vocabria (cabotegravir) 600 mg and long -acting Rekambys (rilpivirine) 900 mg
  Interventions: Drug: Out of Hospital long-acting Vocabria (cabotegravir) 600 mg and long-acting Rekambys (rilpivirine) 900 mg administration

INTERVENTIONS:
Drug: Hospital long-acting Vocabria (cabotegravir) 600 mg and long-acting Rekambys (rilpivirine) 900 mg administration — Hospital administration of long-acting Vocabria (cabotegravir) 600 mg and long-acting Rekambys (rilpivirine) 900 mg as standard of care.
  Other Names: Administration of LA CAB+RPV in the hospital
  Arms: Hospital Group
Drug: Out of Hospital long-acting Vocabria (cabotegravir) 600 mg and long-acting Rekambys (rilpivirine) 900 mg administration — Out of Hospital administration of long-acting Vocabria (cabotegravir) 600 mg and long-acting Rekambys (rilpivirine) 900 mg as an optional therapy in HIV-Infected patients from Spain.
  Other Names: Administration of LA CAB+RPV out of hospital
  Arms: Outpatient Group

SUMMARY:
HOLA is a prospective, randomized (1:1), hybrid type (implementation-effectiveness), phase IV, double arm, open label, multicentric study including virologically suppressed HIVinfected subjects who start or are currently under treatment with the LA antiretroviral combination CAB+RPV, to evaluate the out-of-hospital administration of this combination in terms of acceptability, appropriateness, feasibility and satisfaction.

DETAILED DESCRIPTION:
Randomized patients will receive Long Acting (LA) cabotegravir (CAB) + rilpivirine (RPV) administration in the hospital (standard of care) or out-of-hospital administration every 2 months (M2, M4, M6, M8,M10, M12). Medical visits, routinary blood tests and pharmacy visits at the hospital of reference will take place every 6 months- at baseline, M1 (if patient has not previously receiving LA CAB+RPV), M6 and M12.

ELIGIBILITY:
Inclusion Criteria:

1. Patients equal or older than 18 years old
2. Chronic HIV infection
3. HIV patients in whom LA CAB+RPV is prescribed
4. Recommended triple or dual therapy for at least 12 months, including CAB+RPV LA.
5. Virologically suppression for at least 6 months: 2 consecutive determinations of undetectable viral load (plasma HIV-1 RNA levels < 50 copies/ml ) for ≥ 6 months preceding the study randomization.
6. Post-menopausal or fertile females that agree to avoid pregnancy during the study. If sexually active female; using an effective method of contraception (hormonal contraception, intra-uterine device (IUD), or anatomical sterility in self or partner) from 14 days prior to the first IMP administration until at least 13 months after the last Investigational Medicinal Product (IMP) administration;all female volunteers must be willing to undergo urine pregnancy tests at time points specified in the protocol.
7. Patients which have access to an out of hospital center in which can be treated without inconvenience
8. Patient who agrees to participate in the study and signs the informed consent.

Exclusion Criteria:

1. Hepatitis B infection (section 6.2).
2. History of virological failure or mutations to INSTI or NNRTI.
3. Previous antiretroviral treatment interruption during the last 6 months or treatment interruptions for more than a month.
4. Contraindication for intramuscular injections
5. Pregnancy or breastfeeding women, or with the desire to become pregnant in the near future.
6. Current use of any concomitant treatment as indicated in section 5.6.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the acceptability of the administration of LA CAB + RPV in Alternative Injection Facilities (AOF) from the perspective of participants receiving outside-hospital injections vs the participants receiving hospital injections. | at month 12
  Number of participants receiving injections that show an average composite score ≥ 4 across the AIM questionnaires.
  To asses the acceptability we will use the Acceptability Intervention Measure (AIM) questionnaire (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree). The higher score means the best outcome.
Evaluate the acceptability of the administration of LA CAB + RPV in Alternative Injection Facilities (AOF) from the perspective of participants receiving outside-hospital injections vs the participants receiving hospital injections. | at month 12
  Proportion of participants receiving injections that show an average composite score ≥ 4 across the AIM questionnaires.
  To asses the acceptability we will use the Acceptability Intervention Measure (AIM) questionnaire (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree). The higher score means the best outcome.
Evaluate the acceptability of the administration of LA CAB + RPV in Alternative Injection Facilities (AOF) from the perspective of participants receiving outside-hospital injections vs the participants receiving hospital injections. | at month 12
  Differences among the proportion of participants receiving injections with an average composite score ≥ 4 across the AIM questionnaires.
  To asses the acceptability we will use the Acceptability Intervention Measure (AIM) questionnaire (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree). The higher score means the best outcome.
Evaluate the acceptability of the administration of LA CAB + RPV in Alternative Injection Facilities (AOF) from the perspective of participants receiving outside-hospital injections vs the participants receiving hospital injections. | at month 12
  To asses the acceptability we will use the Acceptability Intervention Measure (AIM) questionnaire (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree). The higher score means the best outcome.
  - Average composite score across the AIM questionnaires.
Assess and compare the CAB + RPV LA - related adverse events (AEs) , all Serious Adverse Events (SAEs), injection site reactions (ISRs) or post injection reactions safety and tolerability of LA CAB+RPV (Safety and Tolerability) | through study completion, an average of 1 year
  Incidence and severity of CAB + RPV LA - related adverse events (AEs) , all Serious Adverse Events (SAEs), Injection site reactions (ISRs) or post injection reactions
Assess and compare the safety and tolerability of LA CAB+RPV. | through study completion, an average of 1 year
  Proportion of participants who discontinue CAB + RPV LA due to AEs/SAEs
Assess and compare the safety and tolerability of LA CAB+RPV. | at month 6 and 12
  Comparing between groups number and proportion of patients who withdraw treatment study due to antiretroviral-related adverse events and reasons
Assess and compare the safety and tolerability of LA CAB+RPV. | at month 6 and 12
  Comparing between groups number and proportion of patients who presented grade 3 or 4 antiretroviral-related adverse events

SECONDARY OUTCOMES:
To assess and compare the acceptability of the administration of LA CAB + RPV as perceived by patients at intermediate times of the study (month 1 and month 6). | at month 1 and 6
  Number of participants receiving injections with an average composite score ≥ 4 across the AIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree) , as perceived by the patient. The higher score means the best outcome.
To assess and compare the acceptability of the administration of LA CAB + RPV as perceived by patients at intermediate times of the study (month 1 and month 6). | at month 1 and 6
  Proportion of participants receiving injections with an average composite score ≥ 4 across the AIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree) , as perceived by the patient.The higher score means the best outcome.
To assess and compare the acceptability of the administration of LA CAB + RPV as perceived by patients at intermediate times of the study (month 1 and month 6). | at month 1 and 6.
  Differences among the proportion of participants receiving injections with an average composite score ≥ 4 across the AIM questionnaires
To assess and compare the acceptability of the administration of LA CAB + RPV as perceived by patients at intermediate times of the study (month 1 and month 6). | at month 1 and 6
  Average composite score across the AIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree) at month 1 and 6. The higher score means the best outcome.
To assess and compare appropriateness and feasibility of the administration of LA CAB + RPV as perceived by patients at month 1, month 6 and month 12. | at months 1, 6 and 12
  Number of participants receiving injections with an average composite score ≥ 4 across the Intervention Appropriateness Measure( IAM) / Feasibility of Intervention Measure (FIM) questionnaires, (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree) as perceived by the patient. The higher score means the best outcome.
To assess and compare appropriateness and feasibility of the administration of LA CAB + RPV as perceived by patients at month 1, month 6 and month 12. | at months 1, 6 and 12
  Proportion of participants receiving injections with an average composite score ≥ 4 across the Intervention Appropriateness Measure( IAM) / Feasibility of Intervention Measure (FIM) questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree), as perceived by the patient.The higher score means the best outcome.
To assess and compare appropriateness and feasibility of the administration of LA CAB + RPV as perceived by patients at month 1, month 6 and month 12. | at month 1, 6 and 12.
  Differences among the proportion of participants receiving injections with an average composite score ≥ 4 across the IAM /FIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree).The higher score means the best outcome.
To assess and compare appropriateness and feasibility of the administration of LA CAB + RPV as perceived by patients at month 1, month 6 and month 12. | at month 1, 6 and 12.
  Average composite score across the Intervention Appropriateness Measure (IAM) and Feasibility Intervention Measure (FIM) patient questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree). The higher score means the best outcome.
To assess and compare the acceptability, appropriateness and feasibility of the administration of LA CAB + RPV as perceived by Healthcare Professionals (HCP)/non-clinical staff at study month 1 and month 6 and month 12. | at months 1, 6 and 12.
  Number of HCP and/or non- clinical staff that show an average composite score ≥ 4 across the Acceptability Intervention Measure (AIM), Intervention Appropriateness Measure (IAM) and Feasibility Intervention Measure (FIM) patient questionnaires questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree).The higher score means the best outcome.
  .
To assess and compare the acceptability, appropriateness and feasibility of the administration of LA CAB + RPV as perceived by Healthcare Professionals (HCP)/non-clinical staff at study month 1 and month 6 and month 12. | at months 1, 6 and 12.
  Proportion of HCP and/or non- clinical staff that show an average composite score ≥ 4 across the AIM / IAM /FIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree).The higher score means the best outcome.
  .
To assess and compare the acceptability, appropriateness and feasibility of the administration of LA CAB + RPV as perceived by HCP/non-clinical staff at study month 1 and month 6 and month 12. | at month 1, 6 and 12.
  Differences among the proportion of HCP/non-clinical staff with an average composite score ≥ 4 across the AIM / IAM /FIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree).The higher score means the best outcome.
To assess and compare the acceptability, appropriateness and feasibility of the administration of LA CAB + RPV as perceived by HCP/non-clinical staff at study month 1 and month 6 and month 12. | at month 1, 6 and 12.
  Average composite score across the AIM / IAM /FIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree).The higher score means the best outcome.
Patient's satisfaction and expectations | baseline and months 1, 6 and 12
  To compare between groups the percentage of patients who report high satisfaction at each study time-points using the HIV Treatment Satisfaction Questionnaire (HIVTSQs12). This scale includes 11 items which are summed to form an 11-item scale score and one item, item 12 (pain/discomfort) is treated as an individual item score.
Patient's satisfaction and expectations | from baseline to months 1, 6 and 12
  To assess changes in satisfaction derived from HIV Treatment Satisfaction Questionnaire status (HIVTSQs12), in the overall sample.
Patient's satisfaction and expectations | from baseline to month 12
  To assess changes in satisfaction derived from HIV Treatment Satisfaction Questionnaire change (HIVTSQc12) in the overall sample.
Patient's satisfaction and expectations | at baseline and month 6 and 12
  To assess and compare among groups the expectations of the LA CAB+RPV regarding the following areas: adherence to treatment, follow-up of medical visits, illness perception, physical and emotional quality of life, family and social relationships and work. Expectations will be assessed through 5-likert scales developed ad hoc for the study
Patient's satisfaction and expectations | baseline and months 1, 6 and 12
  To compare among groups the Patient Reported Outcome Measures (PROMs) at each study time-points using the Patient Reported Outcome Measures HIV Clinic Screening Tool (PROMS-CST- HIV) questionnaire. This questionnaire assesses PRO regarding anticipated stigma, emotional distress, sexuality, social support, material deprivation, sleep and fatigue, cognitive problems, physical symptoms.
Patient's satisfaction and expectations | from baseline to months 1, 6 and 12
  To assess changes in the Patient Reported Outcome Measures (PROMs) throughout the time points in each group in the overall sample using the Patient Reported Outcome Measures HIV Clinic Screening Tool (PROMS-CST- HIV) questionnaire. This questionnaire assesses PRO regarding anticipated stigma, emotional distress, sexuality, social support, material deprivation, sleep and fatigue, cognitive problems, physical symptoms.
Patient's satisfaction and expectations | through study completion, an average of 1 year
  To compare changes in the health professionals 'expectations using a Health Professional Expectations Questionnaire.
Patient's satisfaction and expectations | month 1, 2,4,6,8,10 and month 12.
  To compare the perception of injection, using the perception of injection (PIN) questionnaire.
Retention, engagement and compliance | from baseline to month 6 and 12
  To compare among groups number of patients who miss their appointment for the LA CAB+RPV administration (out of the window period ±7 days)
Retention, engagement and compliance | from baseline to month 6 and 12
  To compare among groups proportion of patients who miss their appointment for the LA CAB+RPV administration (out of the window period ±7 days)
Retention, engagement and compliance | at month 6 and 12.
  To compare among groups number of patients who early interrupt LA CAB+RPV every 2 months
Retention, engagement and compliance | at month 6 and 12.
  To compare among groups proportion of patients who early interrupt LA CAB+RPV every 2 months
Retention, engagement and compliance | at month 6 and 12.
  To compare among groups number of patients who withdraw treatment study
Retention, engagement and compliance | at month 6 and 12.
  To compare among groups proportion of patients who withdraw treatment study
Retention, engagement and compliance | through study completion, an average of 1 year
  Time to LA CAB + RPV discontinuation.
Retention, engagement and compliance | during the 12 months of study.
  To compare among groups the number of patients who adopt oral bridging therapy
Retention, engagement and compliance | during the 12 months of study.
  To compare among groups the proportion of patients who adopt oral bridging therapy
To identify those patients in which the out-of-hospital administration is more suitable. | through study completion, an average of 1 year
  To identify those patients in which the out-of-hospital administration is more suitable by comparing the previous endpoints, stratifying according to: age (< vs >50 years old), gender (male vs female), as well as according to if the participant is already receiving or not LA CAB+RPV.

OTHER OUTCOMES:
To assess and compare between groups the virological effectiveness of CAB + RPV LA | at month 6 and 12.
  Proportion of subjects who are virologically suppressed (plasma HIV-1 RNA ≤ 50 copies/mL)
To assess and compare between groups the virological effectiveness of CAB + RPV LA | at month 6 and 12.
  Proportion of participants with confirmed virologic failure/rebound (2 consecutive HIV-1 RNA greater than or equal to 200 c/mL)
To assess and compare between groups the virological effectiveness of CAB + RPV LA | at month 12
  Proportion of participants with blips
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | from baseline to month 12.
  Difference in number of participants receiving injections that show an average composite score ≥ 4 across the AIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree).The higher score means the best outcome.
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | from baseline to month 12.
  Difference in proportion of participants receiving injections that show an average composite score ≥ 4 across the AIM questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree).The higher score means the best outcome.
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | at month 12
  Average composite score across the Acceptability of Intervention Measure (AIM) questionnaires (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree).The higher score means the best outcome.
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | baseline and month 1, 6 and 12
  To compare between both groups the percentage of patients who report high satisfaction at each study time-points using the Treatment Satisfaction Questionnaire (HIVTSQs12). This scale includes 11 items which are summed to form an 11-item scale score and one item, item 12 (pain/discomfort) is treated as an individual item score.
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | from baseline to month 1, 6 and 12.
  To assess and compare changes in satisfaction derived from HIV Treatment Satisfaction Questionnaire status (HIVTSQs12). This scale includes 11 items which are summed to form an 11-item scale score and one item, item 12 (pain/discomfort) is treated as an individual item score.
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | from baseline to month 12
  To assess and compare changes in satisfaction derived from HIVTSQc12.
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | at baseline and months 6 and 12
  To assess and compare among groups the expectations of the LA CAB+RPV regarding the following areas: adherence to treatment, follow- up of medical visits, illness perception, physical and emotional quality of life, family and social relationships and work. Expectations will be assessed through 5-likert scales developed ad hoc for the study.
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | baseline and months 1, 6 and 12
  To compare among groups the Patient Reported Outcome Measures (PROMs) at each study time-points using the PROMS-CST-HIV questionnaire. This questionnaire assesses PRO regarding anticipated stigma, emotional distress, sexuality, social support, material deprivation, sleep and fatigue, cognitive problems, physical symptoms.
To compare the average change at month 12 vs baseline in patient's acceptability, satisfaction and expectations among the subgroup of participants with previous experience with LA CAB + RPV. | from baseline to months 1, 6 and 12.
  To assess and compare changes in the PROMs throughout the time points in each group.
To compare patient's acceptability, satisfaction and expectations between patients under prior treatment with LA CAB+RPV and those patients who have never received LA CAB+RPV. | at month 12.
  Difference in number and proportion of participants receiving injections that show an average composite score ≥ 4 across the AIM questionnaires.
To compare patient's acceptability, satisfaction and expectations between patients under prior treatment with LA CAB+RPV and those patients who have never received LA CAB+RPV. | at month 12.
  Difference in the average composite score across the Acceptability of Intervention Measure questionnaires (AIM) (item questionnaires that use a 5-point rating scale: 1 = completely disagree to 5 = completely agree). The higher score means the best outcome.
To compare patient's acceptability, satisfaction and expectations between patients under prior treatment with LA CAB+RPV and those patients who have never received LA CAB+RPV. | baseline and month 1, 6 and 12
  To compare between groups the percentage of patients who report high satisfaction at each study time-points using the HIVTSQs12.
To compare patient's acceptability, satisfaction and expectations between patients under prior treatment with LA CAB+RPV and those patients who have never received LA CAB+RPV. | from baseline to month 1, 6 and 12.
  To assess changes in satisfaction derived from HIVTSQs12 .
To compare patient's acceptability, satisfaction and expectations between patients under prior treatment with LA CAB+RPV and those patients who have never received LA CAB+RPV. | from baseline to month 12
  To assess changes in satisfaction derived from HIVTSQc12
To compare patient's acceptability, satisfaction and expectations between patients under prior treatment with LA CAB+RPV and those patients who have never received LA CAB+RPV. | at baseline and months 6 and 12
  To assess and compare among groups the expectations of the LA CAB+RPV regarding the following areas: adherence to treatment, followup of medical visits, illness perception, physical and emotional quality of life, family and social relationships and work. Expectations will be assessed through 5-likert scales developed ad hoc for the study..
To compare patient's acceptability, satisfaction and expectations between patients under prior treatment with LA CAB+RPV and those patients who have never received LA CAB+RPV. | baseline and months 1, 6 and 12
  To compare among groups the PROMs at each study time-points using the PROMS-CST-HIV questionnaire.
To compare patient's acceptability, satisfaction and expectations between patients under prior treatment with LA CAB+RPV and those patients who have never received LA CAB+RPV. | from baseline to months 1, 6 and 12
  To assess changes in the PROMs throughout the time points in each group.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Germans Trias I Pujol Hospital, Badalona, BARCELONA
  - CAP Dr ROBERT, Barcelona, Barcelona
  - Centre de Salut Internacional i Malalties Transmissibles Drassanes - Vall d'Hebron, Barcelona, Barcelona
  - BCN CheckPoint, Barcelona, Barcelona
  - Hospital Vall D' Hebrón, Barcelona, Barcelona
  - Hospital Costa Del Sol, Málaga, Malaga
  - Cs Leganitos, Málaga, Málaga
  - Cs San Pedro de Alcántara, Málaga, Málaga
  - Cs San Luis de Sabinillas, San Luis de Sabinillas, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Processed study data will be in the EU CT Register DB access code 2023-503963-41-00. The raw and personal data protected by privacy laws. After publishing results, the raw dataset that supports the findings of this study are available from sponsor, but data restricted by license, not publicly available. Raw datasets results are, however, available for other researchers from the authors upon reasonable request for collaborative analyses and with the permission of sponsor. Investigators must show the proposed use of the data has been approved by an independent review committee identified for this purpose, and proposal is methodologically sound. Data sharing subject to the regulations (The Organic Law 3/2018 of 5 December on the Protection of Personal Data and the Guarantee of Digital Rights complementary to the Regulation (EU) 2016/679 of 27 April 2016, on protecting individuals regarding processing personal data and free movement).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Final data exportation is scheduled for June 2025 and statistical analyses will follow, with complete datasets expected for the first quarter of 2026.
Access Criteria: Investigators must prove that the proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, and the proposal is methodologically sound. Data sharing is subject to the regulations aforementioned

REFERENCES:
- [Derived] Negredo E, Hernandez-Sanchez D, Alvarez-Lopez P, Falco V, Rivero A, Jusmet J, Cuerda Palomo MA, Flores de la Cruz AB, Pavon JM, Llavero N, Campany D, Faus V, Broto-Cortes C, Bailon L, Aguilar D, Ruiz F, Miranda C, Puig J, Rovira D, Olalla J. Exploring the acceptability, appropriateness, feasibility and satisfaction of an implementation strategy for out-of-HOspital administration of the Long-Acting combination of cabotegravir and rilpivirine as an optional therapy for HIV in Spain (the HOLA study)-a hybrid implementation-effectiveness, phase IV, double-arm, open-label, multicentric study: study protocol. BMJ Open. 2025 Apr 10;15(4):e088514. doi: 10.1136/bmjopen-2024-088514. PMID 40216420